CLINICAL TRIAL: NCT07207564
Title: Integrating Molecular Pathology, Radiology, and Genetics to Improve Breast Cancer Risk
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-009436; NCI-2025-06873 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-009436 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-09-26; First posted 2025-10-06 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Deidentified samples will be stored for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants complete a questionnaire, undergo collection of saliva or blood samples, and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
The purpose of this research is to better understand how benign breast diseases might lead to breast cancer, focusing on genetic factors and including a diverse range of participants to improve future diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, ages 18 to 100 years
* Had a benign breast biopsy at Mayo Clinic between 2002-2022

Exclusion Criteria:

* All male patients
* Prior or concomitant diagnosis of BC
* Diagnosis of BC within six months of benign breast disease
* Denial of research authorization
* Concurrent or post-biopsy bilateral prophylactic mastectomy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who had a benign breast biopsy at Mayo Clinic between 2002 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic features | Baseline (collection of blood or saliva sample)
  Will examine pathologic features from benign tissue to define features related to breast cancer (BC) risk.
Radiologic features | Baseline (collection of blood or saliva sample)
  Will examine radiologic features from mammographic images at time of benign breast disease (BBD) to define features in mammogram images that predict BC risk among women who have a history of BBD. We will also assess whether these features predict BC risk among women without a history of BBD.
Molecular features | Baseline (collection of blood or saliva sample)
  Will examine molecular features to understand how molecular features, including DNA damage and repair work in the breast tissues of women with BBD and how this might relate to risk of developing BC

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Sherman, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No